CLINICAL TRIAL: NCT00044486
Title: A Randomized Controlled Trial of Posaconazole (SCH 56592) vs. Standard Azole Therapy for the Prevention of Invasive Fungal Infections Among High-Risk Neutropenic Patients
Brief Title: Prophylaxis Trial of Posaconazole Versus Standard Azole Therapy for Neutropenic Patients (Study P01899)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P01899
Record Dates: First submitted 2002-08-29; First posted 2002-09-04 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Leukemia, Myelocytic, Acute; Myelodysplastic Syndromes; Neutropenia
Keywords: Prophylaxis; neutropenia; AML; MDS; fungal infections; Acute Myelogenous Leukemia; Anticipated prolonged profound neutropenia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neutropenia; Mycoses

INTERVENTIONS:
Drug: Posaconazole oral suspension

SUMMARY:
This trial is in high risk patients to determine the safety and efficacy of posaconazole vs. fluconazole in the prophylaxis against development of invasive fungal infections.

Profound, prolonged neutropenia (Absolute neutrophil count<500 cells/cubic mm for at least 7 days) due to induction chemotherapy for acute myelogenous leukemia, or myelodysplastic syndrome.

Treatment Duration: maximum of 12 weeks Follow-Up 2 months. Endpoints: incidence of proven or probable IFI according to EORTC/MSG criteria within the neutropenic episode and within 100 days of randomization as determined by external expert review.

DETAILED DESCRIPTION:
This study is designed to determine the safety, tolerance and efficacy of POZ used as prophylaxis if IFI in high-risk subjects with prolonged profound neutropenia. The primary objective is to assess the efficacy of SCH 56592 vs fluconazole and itraconazole in preventing proven or probable IFI during neutropenic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Adults or adolescents (age>13 years) and weight> 34kg, either gender
* Disease definition: Anticipated or documented prolonged neutropenia (ANC<500/mm3 2) Eastern Cooperative Oncology Group (ECOG) performance score of less than 3.
* Female subjects of childbearing age must be using a medically accepted method of birth control before beginning study-drug treatment and agree to continue its use during the study or be surgically sterilized (eg, hysterectomy or tubal ligation).
* Female subjects of childbearing potential must have a negative serum pregnancy test (beta-hcG) at Baseline or within 72 hours before the start of the study drug.

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant, or are nursing.
* Excluded prior treatments: Subjects previously treated with AMB, FLZ, or ITZ for proven or probable IFI within 30 days of enrollment.
* Excluded treatments prior to specific study phases: Subjects who have taken the following drugs: those known to interact with azoles and that may lead to life-threatening side effects.
* Subjects who have used any investigational drugs or biologic agents other than their chemotherapy regimens within 30 days of study entry.
* Subjects who are participating in any other blinded clinical study within 30 days of study entry.
* Subjects with renal insufficiency (estimated creatinine clearance less than 20 mL/minute at Baseline or likely to require dialysis during the study).
* Subjects having an ECG with a prolonged QTc interval by manual reading: QTc greater than 450 msec for men and greater than 470 msec for women.
* Subjects with moderate or severe liver dysfunction at baseline, defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase levels greater than 5 times the upper limit of normal (ULN), or a total bilirubin level greater than 3 times the ULN.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2002-07; Primary Completion 2004-12 (Actual); Study Completion 2005-04 (Actual)

REFERENCES:
- [Derived] Cornely OA, Maertens J, Winston DJ, Perfect J, Ullmann AJ, Walsh TJ, Helfgott D, Holowiecki J, Stockelberg D, Goh YT, Petrini M, Hardalo C, Suresh R, Angulo-Gonzalez D. Posaconazole vs. fluconazole or itraconazole prophylaxis in patients with neutropenia. N Engl J Med. 2007 Jan 25;356(4):348-59. doi: 10.1056/NEJMoa061094. PMID 17251531
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html